CLINICAL TRIAL: NCT04902326
Title: Integrating Behavioral Economics and Self-Determination Theory to Advance Patient Engagement in Diabetes Prevention
Brief Title: Behavioral Economics and Self-Determination Theory to Change Diabetes Risk (BEST Change)
Acronym: BEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jeffrey T. Kullgren, Associate Professor of Internal Medicine and Assistant Professor of Health Management and Policy, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HUM00188543; 1R18DK122418-01 (NIH)
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Pre Diabetes
Keywords: Prevention
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: All investigators, data analysts, and the project manager will be blinded to arm assignment until primary outcome data are collected
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Enhanced Usual Care (EUC) (Active Comparator): Receives one intervention: automated educational text messages
  Interventions: Behavioral: Automated educational text messages
- Financial Incentives (Experimental): Receives two interventions: automated educational text messages and financial incentives.
  Interventions: Behavioral: Automated educational text messages; Behavioral: Financial incentives
- Tailored Messages (Experimental): Receives two interventions: autonomy-supportive automated educational text messages and tailored text messages.
  Interventions: Behavioral: Autonomy-supportive automated educational text messages; Behavioral: Tailored text messages
- Combo Arm-Financial Incentives Plus Tailored Messages Arm (Experimental): Receives three interventions: autonomy-supportive automated educational text messages, tailored text messages, and financial incentives.
  Interventions: Behavioral: Autonomy-supportive automated educational text messages; Behavioral: Financial incentives; Behavioral: Tailored text messages

INTERVENTIONS:
Behavioral: Automated educational text messages — During the first two weeks, participants receive a series of educational messages delivered via text message. These messages welcome participants to the study, set expectations for the next 12 months, and establish a general level of knowledge among all participants on prediabetes, the Diabetes Prevention Program (DPP), and metformin.
  For the next 11.5 months, participants receive three automated text messages per week that provide evidence-based educational content about prediabetes and tips on prevention. Additionally, participants receive monthly messages reminding them about their health insurance plan's coverage of the DPP at no cost and coverage of metformin as a low co-pay medication, and monthly messages providing feedback on their participation in the DPP and use of metformin in the previous calendar month. Participants' PCPs receive quarterly chart updates about participation in the DPP and use of metformin, and A1c results at enrollment and 6 and 12 months.
  Arms: Enhanced Usual Care (EUC); Financial Incentives
Behavioral: Autonomy-supportive automated educational text messages — Participants receive the same text messages as in the automated educational text message intervention, but the thrice weekly messages have been modified, where applicable, to support the participant's autonomy, in accordance with principles of Self-Determination Theory. Participants' PCPs receive quarterly chart updates about participation in the DPP and use of metformin, and A1c results at enrollment and 6 and 12 months.
  Arms: Combo Arm-Financial Incentives Plus Tailored Messages Arm; Tailored Messages
Behavioral: Financial incentives — Participants in this arm have the opportunity to earn a financial incentive ranging from $50 to $250 per month for taking an evidence-based action to prevent T2DM (i.e., engagement in a DPP or fill of a metformin prescription) in the previous month.
  Arms: Combo Arm-Financial Incentives Plus Tailored Messages Arm; Financial Incentives
Behavioral: Tailored text messages — Participants receive twice-weekly tailored text messages that link evidence-based actions to prevent T2DM to the participant's self-identified top values, roles, and strengths. Text messages are also tailored, when possible, to participants' self-reported importance of taking action to try to prevent T2DM (i.e., participating in the DPP or taking metformin), confidence in being able to take such preventive action, and past preventive actions taken.
  Arms: Combo Arm-Financial Incentives Plus Tailored Messages Arm; Tailored Messages

SUMMARY:
Patients with prediabetes can significantly reduce their risk of developing type 2 diabetes mellitus (T2DM) by participating in a Diabetes Prevention Program (DPP) or using metformin, but very few patients with prediabetes engage in these strategies. This randomized controlled trial will compare, among adults with prediabetes, the effectiveness of financial incentives, tailored messages based on self-determination theory (SDT) principles, and the combination of financial incentives plus tailored messages based on SDT principles in decreasing hemoglobin A1c (HbA1c) and weight and in increasing participation in a DPP or use of metformin. Our main hypotheses are that the mean decrease in HbA1c will be greater in the arm that receives a combination of financial incentives plus tailored messages than in the arm that receives generic health education messages, and that the mean decrease in HbA1c will be greater in the arm that receives a combination of financial incentives plus tailored messages than in the arm that receives financial incentives alone and the arm that receives tailored messages alone. The study will also identify moderators and mediators of the effectiveness of the interventions and evaluate facilitators of and barriers to scalability, acceptability, and sustainability of the different interventions.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care Provider part of Michigan Medicine
* Body mass index (BMI) of 25 or higher (23 or higher if of Asian descent)
* Primary health insurance is U-M Premier Care
* Recent Hgb (hemoglobin) A1c 5.7 - 6.4% (inclusive)

Exclusion Criteria:

* Participated in pretesting of intervention materials
* Diagnosis of type 2 Diabetes Mellitus
* Serious mental health conditions (described by protocol)
* End stage renal disease (described by protocol)
* Alcohol dependence and opioid dependence (described by protocol)
* Unable to send and receive several text messages weekly
* No regular access to a smart phone or tablet with data capabilities or Wireless Fidelity (WiFi) connection at home
* Currently taking metformin
* Unable to take metformin due to contraindications or side effects
* Participated in a Diabetes Prevention Program covered by University of Michigan Premier Care insurance
* Currently enrolled in an interventional research study that is examining how a diet, program, or drug might: promote physical exercise, healthy eating habits, or weight loss; lower blood pressure; or lower blood sugar
* Not planning to live in local area over the next year
* Pregnant or planning a pregnancy in the next year
* Received treatment for an eating disorder (e.g. anorexia or bulimia), not including binge-eating disorder, in last 12 months
* Intensive cancer treatment such as bone marrow transplant, chemotherapy, radiation, or cancer related surgery (not including hormonal chemotherapy like Tamoxifen) in last six months or near future
* Organ transplant in last six months
* Bariatric/ gastric bypass surgery, gastric sleeve surgery, or gastric balloon procedure in last six months
* Stroke, heart attack, heart surgery, or hospitalization for congestive heart failure in the past three months
* Other serious health issues or personal concerns that could prevent participant from completing study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kullgren, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data will be made available after conclusion of the study upon written request to the study team and approval of the Principal Investigator.
Supporting Information: Study Protocol, ICF
Time Frame: Once study results are posted on this site (by the primary completion date--no later than 12 months after all primary outcome data have been collected), the de-identified data will be available for five years.
Access Criteria: The de-identified data will be made available after conclusion of the study upon written request to the study team and approval of the Principal Investigator.

REFERENCES:
- [Derived] Carter EW, Vadari HS, Stoll S, Rogers B, Resnicow K, Heisler M, Herman WH, Kim HM, McEwen LN, Volpp KG, Kullgren JT. Study protocol: Behavioral economics and self-determination theory to change diabetes risk (BEST Change). Contemp Clin Trials. 2023 Jan;124:107038. doi: 10.1016/j.cct.2022.107038. Epub 2022 Nov 30. PMID 36460265

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Usual Care (EUC): Receives one intervention: automated educational text messages
  Automated educational text messages: During the first two weeks, participants receive a series of educational messages delivered via text message. These messages welcome participants to the study, set expectations for the next 12 months, and establish a general level of knowledge among all participants on prediabetes, the Diabetes Prevention Program (DPP), and metformin.
  For the next 11.5 months, participants receive three automated text messages per week that provide evidence-based educational content about prediabetes and tips on prevention. Additionally, participants receive monthly messages reminding them about their health insurance plan's coverage of the DPP at no cost and coverage of metformin as a low co-pay medication, and monthly messages providing feedback on their participation in the DPP and use of metformin in the previous calendar month. Participants' PCPs receive quarterly chart updates about participation in the DPP and use of metformin, and A1c results at enrollment and 6 and 12 months.
- Financial Incentives: Receives two interventions: automated educational text messages and financial incentives.
  Automated educational text messages: During the first two weeks, participants receive a series of educational messages delivered via text message. These messages welcome participants to the study, set expectations for the next 12 months, and establish a general level of knowledge among all participants on prediabetes, the Diabetes Prevention Program (DPP), and metformin.
  For the next 11.5 months, participants receive three automated text messages per week that provide evidence-based educational content about prediabetes and tips on prevention. Additionally, participants receive monthly messages reminding them about their health insurance plan's coverage of the DPP at no cost and coverage of metformin as a low co-pay medication, and monthly messages providing feedback on their participation in the DPP and use of metformin in the previous calendar month. Participants' PCPs receive quarterly chart updates about participation in the DPP and use of metformin, and A1c results at enrollment and 6 and 12 months.
  Financial incentives: Participants in this arm have the opportunity to earn a financial incentive ranging from $50 to $250 per month for taking an evidence-based action to prevent T2DM (i.e., engagement in a DPP or fill of a metformin prescription) in the previous month.
Period: Overall Study
Arm/Group | Enhanced Usual Care (EUC) | Financial Incentives | Tailored Messages | Combo Arm-Financial Incentives Plus Tailored Messages Arm
Started | 95 | 95 | 95 | 95
6-month Assessment (Participants who completed at least one of the following three assessments at 6 months: HbA1c, weight, and survey to assess potential mediators and moderators.) | 85 | 88 | 90 | 88
Completed (Participants who completed at least one of the following three assessments at 12 months: HbA1c, weight, and survey to assess potential mediators and moderators.) | 80 | 78 | 81 | 88
Not Completed | 15 | 17 | 14 | 7
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 1
Not completed — Lost to Follow-up | 14 | 14 | 14 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care (EUC) | Tailored Messages | Financial Incentives | Combo Arm-Financial Incentives Plus Tailored Messages Arm | Total
Number analyzed (Participants) | 95 | 95 | 95 | 95 | 380
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (9.7) | 54.2 (9.3) | 53.0 (10.7) | 54.8 (8.7) | 53.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 44 | 63 | 61 | 227
  Male | 36 | 51 | 32 | 34 | 153
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: Non-Hispanic White | 64 | 61 | 65 | 69 | 259
  Race and Ethnicity: Non-Hispanic Black | 15 | 13 | 9 | 13 | 50
  Race and Ethnicity: HIspanic | 3 | 5 | 6 | 2 | 16
  Race and Ethnicity: Other/ mized Non-Hispanic | 13 | 16 | 15 | 11 | 55
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 95 | 95 | 95 | 95 | 380
Education [Count of Participants; unit: Participants]
  4 years or less of college | 58 | 47 | 43 | 54 | 202
  More than 4 years of college | 36 | 48 | 52 | 41 | 177
  Missing | 1 | 0 | 0 | 0 | 1
Income [Count of Participants; unit: Participants]
  Less than $45,000 | 8 | 6 | 8 | 6 | 28
  Greater than and equal to $45,000 | 81 | 83 | 82 | 83 | 329
  missing | 6 | 6 | 5 | 6 | 23
Baseline HbA1c [Mean (Standard Deviation); unit: millimoles per mole (mmol/mol)] | 5.9 (0.2) | 5.9 (0.2) | 5.9 (0.2) | 5.9 (0.2) | 5.9 (0.2)
Baseline weight [Mean (Standard Deviation); unit: pounds] | 217.7 (53.2) | 213.3 (53.2) | 213.9 (49.8) | 199.2 (42.3) | 211.0 (50.1)
Baseline autonomous motivation [Count of Participants; unit: Participants] — Treatment Self-Regulation questionnaire (TSRQ) autonomous motivation sub-scale was summed together and dichotomized at the score of 35, into high and low motivation
  Participants
    High baseline autonomous motivation | 68 | 68 | 68 | 69 | 273
    Low baseline autonomous motivation | 27 | 27 | 27 | 26 | 107

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c From Baseline to 6 Months
Description: Hemoglobin A1C will be tested at a clinical lab using blood samples from venipuncture. An A1C test measures the percentage of red blood cells with glucose-coated hemoglobin. This percentage indicates average blood sugar levels over the last 2-3 months. Higher percentages indicate higher blood sugar levels, and an A1c between 5.7% and 6.4% is considered in the prediabetes range. The negative numbers for change over time indicate an improvement because they show a drop in percentages from the baseline percentages. Changes in HbA1c will be calculated by subtracting the baseline value from the 6-month value, with a negative value indicating an HbA1c reduction.
Time Frame: baseline to 6 months
Population: Data is provided for all individuals who completed an A1c measurement at 6 months. Reported means and confidence intervals are from adjusted models.
Measure: Mean (95% Confidence Interval); unit: percentage of hemoglobin A1c
Arm/Group | Enhanced Usual Care (EUC) | Financial Incentives | Tailored Messages | Combo Arm-Financial Incentives Plus Tailored Messages Arm
Number analyzed (Participants) | 81 | 87 | 89 | 88
percentage of hemoglobin A1c | -0.05 [-0.14 to 0.03] | -0.05 [-0.14 to 0.03] | -0.04 [-0.12 to 0.04] | -0.04 [-0.13 to 0.04]
Statistical Analysis 1: Comparison: Enhanced Usual Care (EUC) vs Financial Incentives vs Tailored Messages vs Combo Arm-Financial Incentives Plus Tailored Messages Arm; Compare the mean decrease of HbA1c of the Combo Arm, Financial Incentives arm, and the Tailored Messages arm each with the EUC arm; Test type: Superiority; p = 0.78, Regression, Linear

2. Primary Outcome: Change in Hemoglobin A1c From Baseline to 12 Months
Description: Hemoglobin A1C will be tested at a clinical lab using blood samples from venipuncture. An A1C test measures the percentage of red blood cells with glucose-coated hemoglobin. This percentage indicates average blood sugar levels over the last 2-3 months. Higher percentages indicate higher blood sugar levels, and an A1c between 5.7% and 6.4% is considered in the prediabetes range. The negative numbers for change over time indicate an improvement because they show a drop in percentages from the baseline percentages. Changes in HbA1c will be calculated by subtracting the baseline value from the 12-month value, with a negative value indicating an HbA1c reduction.
Time Frame: baseline to 12 months
Population: In the combo arm, 5 individuals who completed the study did not complete A1c measurement at 12 months. Reported means and confidence intervals are from adjusted models.
Measure: Mean (95% Confidence Interval); unit: percentage of hemoglobin A1c
Arm/Group | Enhanced Usual Care (EUC) | Financial Incentives | Tailored Messages | Combo Arm-Financial Incentives Plus Tailored Messages Arm
Number analyzed (Participants) | 80 | 78 | 81 | 83
percentage of hemoglobin A1c | -0.14 [-0.25 to -0.03] | -0.10 [-0.21 to 0.01] | -0.12 [-0.22 to 0.00] | -0.12 [-0.23 to 0.00]
Statistical Analysis 1: Comparison: Enhanced Usual Care (EUC) vs Financial Incentives vs Tailored Messages vs Combo Arm-Financial Incentives Plus Tailored Messages Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.64, Regression, Linear

3. Secondary Outcome: Change in Weight From Baseline to 6 Months
Description: Participants will measure their body weight (in pounds) using a scale shipped to them by the study. Participants will submit a photo of the weight displayed on the scale. Change in weight will be calculated by subtracting the baseline value from the 6-month value, with a negative value indicating a weight reduction.
Time Frame: baseline to 6 months
Population: Data is provided for all individuals who sent in their weight at 6 months. Reported means and confidence intervals are from adjusted models.
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Enhanced Usual Care (EUC) | Financial Incentives | Tailored Messages | Combo Arm-Financial Incentives Plus Tailored Messages Arm
Number analyzed (Participants) | 82 | 80 | 85 | 86
pounds | -9.63 [-15.19 to -4.06] | -9.61 [-15.15 to -4.07] | -11.11 [-16.50 to -5.72] | -10.63 [-16.13 to -5.12]
Statistical Analysis 1: Comparison: Enhanced Usual Care (EUC) vs Financial Incentives vs Tailored Messages vs Combo Arm-Financial Incentives Plus Tailored Messages Arm; Compare the mean decrease of weight of the Combo Arm, Financial Incentives arm, and the Tailored Messages arm each with the EUC arm; Test type: Superiority; p = 0.87, Regression, Linear

4. Secondary Outcome: Change in Weight From Baseline to 12 Months
Description: Participants will measure their body weight (in pounds) using a scale shipped to them by the study. Participants will submit a photo of the weight displayed on the scale. Change in weight will be calculated by subtracting the baseline value from the 12-month value, with a negative value indicating a weight reduction.
Time Frame: baseline to 12 months
Population: Data is provided for all individuals who sent in their weight at 12 months. Reported means and confidence intervals are from adjusted models.
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Enhanced Usual Care (EUC) | Financial Incentives | Tailored Messages | Combo Arm-Financial Incentives Plus Tailored Messages Arm
Number analyzed (Participants) | 75 | 72 | 76 | 79
pounds | -10.20 [-17.37 to -3.01] | -8.77 [-15.90 to -1.64] | -10.63 [-17.53 to -3.73] | -11.02 [-18.02 to -4.02]
Statistical Analysis 1: Comparison: Enhanced Usual Care (EUC) vs Financial Incentives vs Tailored Messages vs Combo Arm-Financial Incentives Plus Tailored Messages Arm; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.87, Regression, Linear

5. Secondary Outcome: Engagement in Diabetes Prevention Program or Use of Metformin
Description: Monthly activity of participants enrolled in an online Diabetes Prevention Program (DPP) will be obtained from the program provider. Prescription fills of metformin will be collected from pharmacy benefits data, and proportion days covered (PDC) will be calculated for each month. For months 2-12 a participant is in the study, they will be considered engaged if the calculated metformin PDC for that month was 80% or higher or if they reached the monthly threshold for DPP engagement (4 lessons completed plus at least two of following for at least 4 days: tracked food intake, weighed themselves, and tracked physical activity). Total number of months engaged will be calculated for each participant. Engagement is not assessed in the first month of the study to allow for time to commence engagement.
Time Frame: Months 2-12 of participation in the study
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Enhanced Usual Care (EUC) | Financial Incentives | Tailored Messages | Combo Arm-Financial Incentives Plus Tailored Messages Arm
Number analyzed (Participants) | 95 | 95 | 95 | 95
months | 3.6 (4.2) | 6.6 (4.5) | 4.0 (4.1) | 7.2 (4.1)
Statistical Analysis 1: Comparison: Enhanced Usual Care (EUC) vs Financial Incentives vs Tailored Messages vs Combo Arm-Financial Incentives Plus Tailored Messages Arm; Compare the mean months engaged (with DPP or metformin) of the Combo Arm, Financial Incentives arm, and the Tailored Messages arm each with the EUC arm; Test type: Superiority; p < 0.0001, Regression, Linear

ADVERSE EVENTS:
Time Frame: 12 months for each participant, from randomization to end of study participation
Description: Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Enhanced Usual Care (EUC) | Financial Incentives | Tailored Messages | Combo Arm-Financial Incentives Plus Tailored Messages Arm
All-Cause Mortality (participants affected / at risk) | 0/95 | 1/95 | 0/95 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT04902326/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT04902326/ICF_000.pdf